CLINICAL TRIAL: NCT04614883
Title: Analysis of Volatile Organic Compounds in Exhaled Air and in Sweat in Patients Referred to the Emergency Reception Service for Suspected COVID-19 Infection: Diagnostic Value and for Rapid Screening
Brief Title: Analysis of Volatile Organic Compounds in Exhaled Air and in Sweat in the Context of Suspicion of COVID-19 Infection
Acronym: VOC-COVID-Diag
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_0143
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Asymptomatic patients or Healthy volunteers (Other): Patient with no symptom of COVID-19 infection but for whom a PCR test needs to be done because he has been in contact with a COVID-19 positive person
  Interventions: Device: Volatile Organic Compounds analysis; Other: Canine odor detection of Volatile Organic Compounds
- Symptomatic patients with positive PCR (Other): Patients with symptoms of COVID-19 and whose PCR result is positive
  Interventions: Device: Volatile Organic Compounds analysis; Other: Canine odor detection of Volatile Organic Compounds
- Symptomatic patients with negative PCR but with seroconversion within 4 to 8 weeks (Other): Patients with symptoms of COVID-19 and whose PCR result is negative at inclusion but presents a seroconversion within 4 to 8 weeks post inclusion
  Interventions: Device: Volatile Organic Compounds analysis; Other: Canine odor detection of Volatile Organic Compounds

INTERVENTIONS:
Device: Volatile Organic Compounds analysis — VOC analysis in exhaled air with e-noses and mass spectrometry. VOC analysis in sweat with mass spectrometry.
Other: Canine odor detection of Volatile Organic Compounds — VOC analysis in sweat by trained dogs.

SUMMARY:
In the context of the actual pandemia of the Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) which requires a better diagnostic strategy for the management of patients.

The study of volatile organic compounds (VOC) detected in exhaled air or in sweat, is an innovative research area for respiratory diseases. The analysis of VOC can be done either by the technique of the mass spectrometry which allows the identification of each VOC in the exhaled air or by the technique of electronic nose, simpler and faster, which provides an idea of the general profile of the VOC without identifying them. The VOC have shown their interest in some situations, such as diagnostic or prognostic tool in patients followed for thoracic tumorous pathology or bronchial or pulmonary vascular diseases.

Moreover, it has recently been shown that properly trained dogs would be able to detect an olfactory signature of SARS-CoV-2 infection with a specificity greater than 90%; this olfactory signature corresponds to VOCs detectable by the flair of dogs (Nosaïs-Covid19 study).

Validation of the diagnostic value of VOC analyzes by non-invasive and rapid methods (electronic nose analysis or mass spectrometry; detection by the scent of dogs) for the rapid detection and early diagnosis of a SARS-CoV-2 infection warrants the performance of this clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients

   * Patents anaged at the Foch Hospital for suspected COVID-19 and any other patient whose management requires diagnosis of SARS-CoV-2 infection
   * Patients aged 18 or over;
   * Patients Fluent in French ;
   * Patients with a signed consent form;
   * Patients with a health insurance plan.
2. Healthy volunteers

   * Foch Hospital staff asymptomatic for SARS-CoV-2 infection;
   * Aged 18 yor over;
   * Fluent in french;
   * with a signed consent form;
   * With a health insurance plan.

Exclusion Criteria:

* Pregnant woman
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Validate the interest of VOCs analyzed by electronic noses and / or mass spectrometry for the diagnosis of a COVID-19 infection | 1 day
  Comparison of variation of Volatile Organic Compound (VOC) profiles in exhaled air of patients between patients with symptoms suggestive of COVID and infection confirmed by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) and those whose infection is ruled out based on the negativity of RT-PCR and clinical data

SECONDARY OUTCOMES:
Identify the nature of VOCs associated with infection by SARS-CoV-2 by mass spectrometry in exhaled air and in sweat | 1 day
  The equivalences and differences in nature of VOCs associated with infection with SARS-CoV-2 between exhaled air and sweat.
Assessment of the specificity and sensitivity of canine olfactory detection of COVs associated with infection by SARS-CoV-2 (COVID-19) | 1 day
  Proportion of success in detecting samples from patients with symptoms suggestive of COVID and infection confirmed by PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Salvator, MD, Principal Investigator — Hopital Foch
Locations (1):
- Foch hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No